CLINICAL TRIAL: NCT07111065
Title: Phase II, Randomized, Double-Blind, Placebo-Controlled Trial of Omega-3 Fatty Acid (O3FA) Supplementation for Adult and Juvenile Dermatomyositis (DM/JDM)
Brief Title: FAST for DM Fatty Acid Supplementation Trial (FAST) for Dermatomyositis (DM)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10001790; 001790-E
Record Dates: First submitted 2025-08-07; First posted 2025-08-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-26

CONDITIONS: Dermatomyositis (DM); Juvenile Dermatomyositis (JDM)
Keywords: Fish oil supplements; Omega-3 Fatty Acid; Dietary Guidelines for Americans; Clinical Trial; Online questionnaires; Diet Study
MeSH Terms: conditions — Dermatomyositis | interventions — Fish Oils; Nutrition Policy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 Fatty Acid Fish Oil Dietary Supplement and Dietary Guidelines for Americans diet (Active Comparator): Fish oil supplement and healthy diet
  Interventions: Dietary Supplement: FISH OIL 500MG OMEGA-3 SOFT GEL MINIS; Other: Dietary Guidelines for Americans diet
- Placebo and Dietary Guidelines for Americans diet (Placebo Comparator): Placebo capsules look identical to fish oil but contain corn oil, complemented by healthy diet
  Interventions: Other: Dietary Guidelines for Americans diet

INTERVENTIONS:
Dietary Supplement: FISH OIL 500MG OMEGA-3 SOFT GEL MINIS — Translucent, light yellow, oblong soft gelatin capsule containing a straw to amber light liquid.
  Arms: Omega-3 Fatty Acid Fish Oil Dietary Supplement and Dietary Guidelines for Americans diet
Other: Dietary Guidelines for Americans diet — The Dietary Guidelines provides science-based advice on what to eat and drink to promote health, help reduce risk of chronic disease, and meet nutrient needs.

SUMMARY:
Dermatomyositis (DM) is a rare autoimmune disease that causes muscle weakness, skin rashes, and other symptoms. Researchers think both genetic and environmental factors play a role in this disease. They want to find out more about how diet and lifestyle choices affect people with DM/JDM.

Objective:

To see if omega-3 fatty acid supplements from fish oil, combined with a healthy diet, can help people with DM/JDM.

Eligibility:

Adults 18-60 years old, who live in the United States, can read English, and access Internet to complete questionnaires can participate.

Design:

Participants will have 5 or 6 inpatient visits. For 5 visits they may need to stay in the Clinical Center for up to 5 days. Participants will be screened. They will have a physical exam with blood, urine and stool tests. They will have tests of their heart and lung function. Their muscle strength will be measured. They may have an imaging scan of their thighs and pelvis. They will complete online questionnaires about their health and lifestyle. They may complete two optional skin biopsies. Participants will take 4 small capsules by mouth twice a day for up to 6 months. The capsules will contain omega-3 fatty acids from fish oil or a placebo. The placebo looks just like the regular capsule but contains no active ingredients. Participants will not know which capsules they are taking. They will follow a healthy diet based on the Dietary Guidelines for Americans.

Participants will receive dietary coaching and will have virtual check-ins throughout the study. For two 7-day periods, they will wear a watch-like device to track their daily activity and sleep patterns. Participants may opt to remain in the study for an additional 12 weeks. All will receive the fish oil supplements during this stage.

DETAILED DESCRIPTION:
Study Description:

Multi-site, randomized, double-blind, placebo-controlled trial to evaluate the efficacy of O3FA supplementation on improving myositis disease activity, including muscle strength and function and other elements of disease activity, and quality of life in patients with mild to moderately active Dermatomyositis (DM)/Juvenile Dermatomyositis (JDM).

Objectives:

Primary Objective:

-To examine the effect of O3FA supplementation on disease activity in a randomized, placebo-controlled trial in patients with mild to moderately active DM/JDM.

Secondary Objectives:

* To examine the effect of O3FA supplementation on DM/JDM disease activity.
* To assess the safety and tolerability of O3FA supplementation in patients with DM/JDM.

Exploratory Objectives:

* To examine the effects of O3FA supplementation on measures of muscle strength and function, patient reported outcomes, vascular/endothelial function, mediators of inflammation and autoimmunity and other measures of DM/JDM disease activity
* To examine effects of O3FAs on metabolic parameters and lipids
* To examine the feasibility and compliance with a diet following the Dietary Guidelines for Americans.
* To evaluate the effect of O3FAs and diet following the Dietary Guidelines for Americans on stool microbial diversity.
* To examine the effect of other lifestyle and environmental factors on the O3FA intervention response.

Endpoints:

Primary:

Reduction in DM/JDM disease activity, as assessed by the American College of Rheumatology-European League Against Rheumatism (ACR-EULAR) Myositis Response Criteria Total Improvement Score (TIS), a composite of change in myositis core set activity measures, from Week 0 to Week 24.

Secondary:

Minimum improvement, as defined by ACR-EULAR myositis response criteria (i.e., improvement >= 20 points in the TIS) and change in core set measures of myositis disease activity between week 0 and week 24 and between weeks 0 and 12. Frequency of adverse events (AE) in O3FA vs. Placebo group from week 0 to 24.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Adults 18-60 years of age with probable or definite EULAR-ACR criteria for adult or juvenile dermatomyositis (DM, JDM).
* Willingness to adhere to Dietary Guidelines for Americans dietary regimen, undergo dietary coaching on weekly to biweekly basis (10 sessions), and to complete online random reporting of dietary intake over a 6-month period.
* Ability and willingness to comply with taking 4 study pills twice a day for 6 months.
* Ability and willingness to wear ActiGraph device at home for 7 continuous days, twice in the study.
* Willingness and ability to complete and consent to study testing, including blood, stool, and urine samples, and imaging studies.
* Ability and willingness to complete a total of 5 study visits (screening, weeks-6, 0, 12, 24) onsite at NIH Clinical Center in Bethesda, Maryland.
* Has the ability/transportation methods to attend on-site visits. Willing to pay for travel and out-of-pocket expenses.
* Own or have reliable access to a computer, laptop or smart phone device (iPhone or Android) with internet access, and an active email address, to complete study consent form, online questionnaires, telehealth visits, and review online dietary education materials and videos.
* Ambulatory
* Must live within the United States.
* Must read English (at least 4th grade level) and complete questionnaires in English (forms validated in English). Ability and willingness to complete forms online.
* Moderately active DM/JDM defined by:

  * MD global VAS with a >= 2.0 cm on a 10 cm scale and maximum value of 7.0 cm, and
  * At least 2 of the following criteria:

    * Patient global activity >= 2 cm out of 10 cm visual analog scale (VAS).
    * MMT-8 score of <=138 out of 150.
    * Health Assessment Questionnaire disability index with a minimum value of >= 0.50 out of 3.0
    * Elevation of at least one of the muscle enzymes (which includes creatine kinase (CK), aldolase, lactate dehydrogenase (LDH), ALT and AST) at a minimum level of 1.3X the upper limit of normal.
    * Global Extramuscular disease activity score with a minimum value of >= 1.0 cm on a 10 cm VAS scale (this measure is the physician s composite evaluation and is based on assessments of activity scores on the constitutional, cutaneous, skeletal, gastrointestinal, pulmonary and cardiac scales of the Myositis Disease Activity Assessment Tool (MDAAT).
* Physician global damage and muscle damage both <= 5.0 cm/10 cm VAS
* If receiving prednisone and methotrexate, the dose must be stable for at least 4 weeks prior to the Week-6 visit, and daily prednisone <= 20 mg/day.
* Background therapy with other non-corticosteroid immunosuppressive agent, if required, must be at a stable dose for at least 6 weeks prior to the Week-6 visit, except with IVIG regimen should be stable 90 days prior to the Week-6 visit and for rituximab, stable regimen for 4 months prior to screening Week-6.
* If an immunosuppressive agent was discontinued prior to the screening visit, then there must be a washout period before week-6 visit:

  * 4-week washout for prednisone, methotrexate, and IV methylprednisolone (IV pulse therapy)
  * 8-week washout for other immunosuppressive drugs, including azathioprine, mycophenolate mofetil, leflunomide, tacrolimus, cyclosporine, cyclophosphamide, colchicine, and hydroxychloroquine
  * 8-week washout for IVIG
  * For discontinuation of biologic or targeted drug therapies or dietary supplements, a washout prior to visit 1 (week-6) is required of 4 terminal half-lives.
* Negative pregnancy test (urine or blood sample) if born female.
* Body Mass Index (BMI) > 18 and <= 35 kg/m^2
* Fish intake of less than 2 servings per week on average for the past 3 months.
* Intake of meat products (beef, lamb, pork, venison, rabbit, cow s milk or dairy products) within 2 months of screening visit and of week 0 and have no reaction (no shortness of breath, hives, rash, or diarrhea) within 6 hours of ingestion of these meat products.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Polymyositis; inclusion body myositis; cancer-associated myositis, defined as the diagnosis of myositis within 3 years of the diagnosis of cancer, except basal or squamous cell skin cancer or carcinoma in situ of the cervix if at least 5 years since excision.
* Myositis in overlap with another connective tissue disease (CTD), including overlap with inflammatory bowel disease (Crohn s disease, ulcerative colitis, celiac disease), except patients with overlap of autoimmune thyroid disease (Hashimoto s, Grave s Disease etc.) that is stable and controlled, with no changes in medications over the past 3 months, will be allowed.
* Drug- or toxin-induced myositis, including known HMG-CoA reductase autoantibody-positive necrotizing myopathy following statin use.
* Moderate to severely active myositis that would require initiation of another immunosuppressive treatment.
* Joint disease, severe calcinosis, or other musculoskeletal condition, which precludes the ability to assess/quantitate muscle strength and function.
* Concomitant illness that would prevent adequate patient assessment or in the investigators opinion pose an added risk for study participants. The investigator may consider further evaluation or consultation if clinically indicated prior to study enrollment:

  * Recurrent or chronic infections, including HIV, hepatitis B and C, Epstein Barr virus, active coronavirus infection, active or recurrent gastrointestinal infection (including Helicobacter pylori), active or recurrent skin infections with calcinosis.
  * Disorders that would preclude accurate assessment of neuromuscular function.
  * Severe swallowing dysfunction with inability to swallow pills.
  * Patients with generalized lipodystrophy.
  * Severe cardiomyopathy or arrhythmias, including atrial fibrillation or atrial flutter, New York Heart Association Classification III or IV for congestive heart failure, severe interstitial lung requiring oxygen therapy, gastrointestinal vasculopathy/ulceration or gastroparesis, renal failure requiring dialysis, that in the investigators opinion poses an additional risk for study participants.
  * Subjects with any acute and life-threatening condition unrelated to myositis, such as prior sudden cardiac arrest, acute myocardial infarction, stroke, embolism in last 3 months.
  * History of malignancy, except basal or squamous cell skin cancer or carcinoma in situ of the cervix if at least 5 years since excision.
  * Uncontrolled hypertension with average blood pressure >= 140/90, requiring a new anti-hypertensive medication in the past 8 weeks.
  * Psychiatric illness that precludes compliance or neuromuscular assessment, including major psychiatric illness requiring hospitalization within the past year and/or has had a change in depression or anxiety prescription medications within the past 3 months (by discretion of study physician).
  * Subjects with chronic diarrhea, gastric bypass or lap-band procedures, ostomies, bowel motility problems, irritable bowel syndrome, symptomatic gallstones, or other conditions that could affect intestinal fat absorption.
  * Subjects with clinically diagnosed hepatic disease, including but not limited to hepatitis, steatosis, cirrhosis.
  * Osteoporotic fracture under therapy for pain control or impacting ambulation.
  * Serum creatinine > 2.0mg/dl or eGFR less than 50 mL/min per 1.73 m^2.
  * Subjects with coagulation or bleeding disorders (such as hemophilia) or receiving anti-platelet or anti-coagulant medications, including daily aspirin, warfarin, or Plavix.
  * Life-threatening non-myositis illness that would interfere with the patient s ability to complete the study.
* Known contraindications to O3FAs, excipients or placebo contents (e.g., allergy or known hypersensitivity to that drug or its excipients, including porcine gelatin, allergies to fish or shellfish, tocopherols, glycerin, or corn). Religious or ethical reasons to not consume fish, corn and/or porcine (pork) products.
* Participants with any of the following:

  * Idiopathic anaphylaxis
  * Alpha-gal reaction
  * Known food allergies to beef, pork, lamb or other meat products, including cow s milk and dairy products, with a history of shortness of breath, rash, or hives within 6 hours of eating these foods.
* Currently using O3FAs or consuming EPA/DHA in any form for the past 6 months.
* Currently taking supplements or medications that affect lipoproteins for the past 6 months, including fish oil supplements, bile-acid sequestrants, plant sterol supplements, PCSK9 inhibitors, fibrates, statins, or niacin.
* Use of medications or dietary supplements that interact with O3FA per pharmacy evaluation. A PharmD will evaluate the patient's current medication list for medications/supplements with the potential for significant interactions with O3FA.
* No antibiotic usage in past 3 months, as well as no usage of anti-virals, antifungals, anti-parasitics in past 3 months (except antimalarials and Paxlovid or other COVID-19 anti-viral therapy allowed).
* Subjects being treated with tamoxifen, estrogens or progestins that have not been stable for > 4 weeks.
* Uncontrolled diabetes with HgbA1C > 8 or hospitalization in past 6 months for diabetes.
* Uncontrolled hyperlipidemia with TC > 400 mg/dL, TG >150mg/dL.
* Currently on a weight-loss program
* Has experienced a weight change (gain or loss) of greater than 15 pounds or greater than 20 percent in the past 3 months
* Currently taking a GLP-1 receptor agonist medication
* No restrictive dietary habits per discretion of the study team.
* Current use of medications or dietary supplements for weight or appetite control, including laxatives or diarrheal inhibitors within the past 4 weeks.
* History of eating disorder.
* Initiation of an exercise program within 4 weeks of screening visit.
* Known or suspected history of drug or alcohol abuse within the past 6 months as determined by the medical record or patient interview.
* Blood donation in the last 6 weeks or planned blood donation during study or requiring regular blood transfusion.
* Pregnant females or nursing mothers within past 3 months, or those planning to get pregnant during the next 9 months.
* Low total WBC < 2000, platelets < 100,000/mm3; hemoglobin < 9.5 gm/dl.
* Vitamin D level < 20 ng/ml (at screening visit - necessitates addition of supplement and re-screen after minimum of 8 weeks).
* Subjects with TSH levels greater than 1.5X upper limit of normal or clinical evidence of hypothyroidism (at screening visit- necessitates addition of supplement and re-screen after minimum of 8 weeks).
* Participants with severe claustrophobia.
* History of or anticipated poor non-cooperation with study requirements.
* Participation in another clinical experimental therapeutic study within 30 days of screening visit or during the study.
* Hospitalization within past 30 days (other than for routine infusions).
* Prisoners or subjects who are involuntarily incarcerated.
* Resident of a nursing home, ward of the state, or institutionalized during any part of the study period.
* Persons with decisional incapacity/cognitive impairment.
* Any history or evidence of severe illness or any other condition that would make the patient, in the opinion of the investigator, unsuitable for the study.
* Participants who do not complete the ASA24 within 4 calendar days of screening will be excluded from the protocol. Additionally, participants will be excluded if their energy intake from the ASA24 is above or below established cut-off values for age and gender.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-11-03 (Estimated); Study Completion 2031-11-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in DM/JDM disease activity, as assessed by the ACR-EULAR Myositis Response Criteria Total Improvement Score, a composite assessment of change in myositis core set activity measures, between the O3FA vs. placebo groups. | From Week 0 to Week 24
  Assessed at 24 weeks for the treatment arm (O3FA) and the placebo arm.

SECONDARY OUTCOMES:
Meeting minimum clinical improvement in disease activity in O3FA and placebo groups | From Week 0 to Week 24
  Minimum clinical improvement defined by ACR-EULAR myositis response criteria: improvement of (Bullet) 20 points in the Total Improvement Score (TIS) between the O3FA vs. placebo groups at Week 24
The effects of O3FA on DM/JDM disease activity | From Week 0 to Week 24
  Change in myositis disease activity as assessed by specific core set disease activity measures between the O3FA vs. placebo groups
Safety and Tolerability | From Week 0 to Week 24
  Incidence of adverse events by NCI CTC Adverse Event assessments between the O3FA vs. placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa G Rider, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Participants will be enrolled from a rare disease population, and there is a risk of deidentifying the data.

REFERENCES:
- [Background] Rider LG, Aggarwal R, Machado PM, Hogrel JY, Reed AM, Christopher-Stine L, Ruperto N. Update on outcome assessment in myositis. Nat Rev Rheumatol. 2018 May;14(5):303-318. doi: 10.1038/nrrheum.2018.33. Epub 2018 Apr 12. PMID 29651119
- [Background] Ward JM, Ambatipudi M, O'Hanlon TP, Smith MA, de Los Reyes M, Schiffenbauer A, Rahman S, Zerrouki K, Miller FW, Sanjuan MA, Li JL, Casey KA, Rider LG. Shared and Distinctive Transcriptomic and Proteomic Pathways in Adult and Juvenile Dermatomyositis. Arthritis Rheumatol. 2023 Nov;75(11):2014-2026. doi: 10.1002/art.42615. Epub 2023 Aug 13. PMID 37229703
- [Background] Saygin D, Kim H, Douglas C, Erman B, Wilkerson J, McGrath JA, Oddis CV, Lundberg IE, Amato AA, Garcia-De La Torre I, Chinoy H, Fiorentino D, Chung L, Song YW, Miller FW, Ruperto N, Vencovsky J, Aggarwal R, Rider LG; International Myositis Assessment and Clinical Studies Group (IMACS). Performance of the 2016 ACR-EULAR Myositis Response Criteria in adult dermatomyositis/polymyositis therapeutic trials and consensus profiles. Rheumatology (Oxford). 2023 Nov 2;62(11):3672-3679. doi: 10.1093/rheumatology/kead110. PMID 36929923
- [Background] Tedeschi SK, Costenbader KH. Is There a Role for Diet in the Therapy of Rheumatoid Arthritis? Curr Rheumatol Rep. 2016 May;18(5):23. doi: 10.1007/s11926-016-0575-y. PMID 27032786
- [Background] Gioxari A, Kaliora AC, Marantidou F, Panagiotakos DP. Intake of omega-3 polyunsaturated fatty acids in patients with rheumatoid arthritis: A systematic review and meta-analysis. Nutrition. 2018 Jan;45:114-124.e4. doi: 10.1016/j.nut.2017.06.023. Epub 2017 Jul 8. PMID 28965775
- [Background] Ramessar N, Borad A, Schlesinger N. The effect of Omega-3 fatty acid supplementation in systemic lupus erythematosus patients: A systematic review. Lupus. 2022 Mar;31(3):287-296. doi: 10.1177/09612033211067985. Epub 2022 Jan 13. PMID 35023407
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001790-E.html